CLINICAL TRIAL: NCT05635656
Title: Digital Symptom Mapping and Home-based Biofeedback Treatment for Adults with Persistent Postconcussion Symptoms: a Development and Usability Study
Brief Title: Digital Solutions for Concussion
Acronym: DiSCo
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Olavs Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 422538
Record Dates: First submitted 2022-11-02; First posted 2022-12-02 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2023-04

CONDITIONS: Post-Concussion Syndrome; Post-Traumatic Headache
MeSH Terms: conditions — Post-Concussion Syndrome; Post-Traumatic Headache

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Digital symptom mapping and biofeedback treatment (Experimental)
  Interventions: Device: Digital symptom mapping and biofeedback treatment

INTERVENTIONS:
Device: Digital symptom mapping and biofeedback treatment — Digital symptom mapping and biofeedback treatment

SUMMARY:
The objective of this study is to develop new digital solutions for patients with prolonged postconcussion symptoms, and investigate its usability, feasibility, and safety. The digital solutions consist of a 1) symptom mapping and clinical decision support system, and 2) a research-based system for home-based biofeedback treatment.

ELIGIBILITY:
Inclusion Criteria:

* 18 or older at the time of inclusion.
* Mild TBI as defined by having sustained a head injury with observed or self-reported alteration of consciousness, amnesia, or other relevant acute symptoms.
* PPCS according to the ICD-10 research criteria and PTH according to International Classification of Headache Disorders 3rd edition (ICHD-3). Operationalized as reporting 3 or more symptoms (including headache) on a moderate or greater intensity level on the RPSQ.
* Proficient in Norwegian language (oral and written)
* Signed informed consent

Exclusion Criteria:

* Serious psychiatric or somatic disease, or other patient-related factors, that based on an evaluation of the study personnel responsible for inclusion, will provide obvious challenges for adhering to the protocol, including using the devices.
* Less than three months of experience with smartphones
* Not having access to an iOS or Android smartphone

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2022-11-25 (Actual); Primary Completion 2024-03-05 (Actual); Study Completion 2024-03-05 (Actual)

PRIMARY OUTCOMES:
Usability of new digital solutions for symptom mapping and home-based biofeedback treatment in patients with PPCS/PTH | Will be assessed at three different time points: After each usability testing during the iterative development cycles (T1 and T2) and after the home-testing period (T3).
  - Description mHealth App Usability Questionnaire scores in the target user group; and Mobile App Rating Scale scores by an independent group of clinicians and researchers

SECONDARY OUTCOMES:
Feasibility and adherence of new digital solutions | Will be assessed after the home-testing period (T3)
  * Number of days with logged symptom data during a 4-week home-testing period
  * Number of biofeedback sessions and mean change in biofeedback scores throughout the testing period

OTHER OUTCOMES:
Safety of new digital solutions | Will be assessed at three different time points: After each usability testing during the iterative development cycles (T1 and T2) and after the home-testing period (T3).
  Description of the frequency and severity of adverse events, serious adverse events and unexpected serious adverse events

CONTACTS AND LOCATIONS:
Locations (1):
- St. Olavs Hospital, Trondheim, Norway

IPD SHARING:
Plan to Share IPD: No